CLINICAL TRIAL: NCT02183571
Title: Bioequivalence of Two Strengths (1000 mg and 500 mg) of Two Different Metformin Tablets Administered to Healthy Male and Female Subjects in an Open, Randomised, Single-dose, Two-period Crossover, Phase I Trial
Brief Title: Bioequivalence Study of Two Strengths of Two Different Metformin Tablets Administered to Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.57
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- Glucophage® high dose (Experimental): Part I: Treatment A + B
  Interventions: Drug: Merck Glucophage® high dose; Drug: BMS Glucophage® high dose
- Glucophage® low dose (Experimental): Part II: Treatment C+ D
  Interventions: Drug: Merck Glucophage® low dose; Drug: BMS Glucophage® low dose

INTERVENTIONS:
Drug: Merck Glucophage® high dose — Part I: Treatment A
  Arms: Glucophage® high dose
Drug: BMS Glucophage® high dose — Part I: Treatment B
  Arms: Glucophage® high dose
Drug: Merck Glucophage® low dose — Part II: Treatment C
  Arms: Glucophage® low dose
Drug: BMS Glucophage® low dose — Part II: Treatment D
  Arms: Glucophage® low dose

SUMMARY:
Investigation of bioequivalence of BMS Glucophage® tablets and Merck Glucophage® tablets in the strengths of 1000 mg (part I) and 500 mg (part II)

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG) and clinical laboratory tests
* Age ≥ 18 and Age ≤ 55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination deviating from normal and of clinical relevance. Repeated measurement of a systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration except if a relevant interaction can be ruled out
* Participation in another trial with an investigational drug within two months prior to first study drug administration
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to the start of study)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsade de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

For female subjects:

* Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 1 month after study completion
* No adequate contraception during the study and until 1 month after study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, IUD (intrauterine device), sexual abstinence for at least 1 month prior to enrolment, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who do not have a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to use an additional barrier method (e.g. condom, diaphragm with spermicide)
* Lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity) | up to 48 h after drug administration
Cmax (maximum measured concentration of metformin in plasma) | up to 48 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of metformin in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 48 h after drug administration
AUCt1-t2 (Area under the concentration time curve of metformin in plasma over the time interval t1 to t2) | up to 48 h after drug administration
tmax (time from dosing to the maximum concentration of metformin in plasma) | up to 48 h after drug administration
λz (terminal rate constant in plasma) | up to 48 h after drug administration
t1/2 (terminal half-life of metformin in plasma) | up to 48 h after drug administration
MRTpo (mean residence time of metformin in the body after po administration) | up to 48 h after drug administration
CL/F (apparent clearance of metformin in the plasma after extravascular administration) | up to 48 h after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 48 h after drug administration
Number of patients with clinically relevant differences in physical examination | Baseline, day 1 prior, within 2-10 days following the last study drug administration
Number of patients with clinically relevant differences in vital signs (BP (Blood pressure), PR (Pulse rate)) | Baseline, day 1 prior, within 2-10 days following the last study drug administration
Number of patients with clinically relevant differences in 12-lead ECG (electrocardiogram) | Baseline, day 1 prior, within 2-10 days following the last study drug administration
Number of patients with clinically relevant differences in clinical laboratory tests | Baseline, day 1 prior, within 2-10 days following the last study drug administration
Number of patients with adverse events | within 2- 10 after last study drug administration
Assessment of tolerability by investigator on a 4 point scale | within 2- 10 after last study drug administration